CLINICAL TRIAL: NCT04298112
Title: PSMA-PET and MRI for Detection of Recurrent Prostate Cancer After Radical Treatment - a Multicenter Study
Brief Title: PSMA-PET and MRI for Detection of Recurrent Prostate Cancer After Radical Treatment
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Haukeland University Hospital (Other); University Hospital of North Norway (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 83009
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-04

CONDITIONS: Prostatic Neoplasms
Keywords: Diagnostic Imaging; Positron-Emission Tomography; Magnetic Resonance Imaging; Prostate-Specific Antigen; Neoplasm Recurrence, Local
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Recurrence, Local

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- relapse after radical treatment for prostate cancer: prostate cancer patients with biochemical relapse following radical treatment, or patients with persistently elevated PSA levels after radical prostatectomy, that have been (or will be) referred to PSMA PET/CT and PSMA PET/MRI at one of the participating hospitals.
  Interventions: Diagnostic Test: PSMA PET/CT; Diagnostic Test: PSMA PET/MR

INTERVENTIONS:
Diagnostic Test: PSMA PET/CT — Whole-body PET/CT (contrast enhanced CT or low-dose CT); from vertex to thighs.
Diagnostic Test: PSMA PET/MR — Pelvic PET/MR in addition to targeted PET/MR according to other findings from the PET/CT (e.g. columna)

SUMMARY:
Approximately one third of prostate cancer patients experience biochemical relapse following initial radical prostatectomy or curative radiotherapy. To determine further treatment, it is of utmost importance to accurately differentiate local and regional recurrence from distant metastatic disease. Unfortunately, the currently used medical imaging methods (MRI and bone scan) lack sensitivity for detection of nodal and skeletal metastases, which can lead to over-treatment of patients with occult metastatic disease. PET imaging with prostate specific membrane antigen (PSMA)-ligands has shown a promising potential for improving the detection accuracy in recurrent prostate cancer, especially when combined with the excellent soft-tissue contrast of MRI. However, evidence is mostly based on retrospective single center studies so far, including patients with a wide variety of PSA levels.

Improving the sensitivity for detection of metastatic disease is a crucial step in reducing over-treatment of prostate cancer patients with biochemical relapse following radical treatment. The purpose of this prospective multi-center study is to standardize PSMA PET/CT and PET/MRI imaging across three university hospitals in Norway, and investigate its merit for detection of recurrent prostate cancer. The long-term overall goal is offering prostate cancer patients a more personalized treatment plan aiming to improve the chances of survival and quality of life.

ELIGIBILITY:
Inclusion Criteria (surgery cohort):

* Prostate cancer patients with biochemical relapse in accordance with the European Association of Urology (EAU) guidelines on prostate cancer; two consecutive measurements with PSA ≥ 0.2 ng/ml following radical prostatectomy or PSA > 2.0 ng/ml above the nadir following definitive radiotherapy
* Potential candidates for loco-regional pelvic salvage treatment based on age and co-morbidity

Exclusion Criteria:

* Previous salvage therapy for recurrent prostate cancer
* General contra-indications for an MRI exam (pacemaker, aneurysm clips, any form of metal in the body, or severe claustrophobia)
* Serious concomitant systemic disorders or reduced cognitive functioning that in the opinion of the investigator would compromise the patient's ability to complete the study or interfere with the evaluation of the efficacy and safety of the study objectives
* Impaired renal function defined as estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73 m2
* Hormonal treatment during the last three months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer patients with biochemical relapse after radical treatment, or patients with persistently elevated PSA levels after radical prostatectomy, who have been (or will be) referred to standardized PSMA PET/CT and PSMA PET/MRI at one of the participating Norwegian hospitals.
  Based on the local patient populations, 120 patients are expected to be included in Trondheim, 120 in Bergen, and 60 in Tromsø.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Detection rates of prostate cancer recurrence after radical treatment using a standardized imaging protocol consisting of PSMA PET/CT and PET/MR | baseline
  Consensus scoring and decision by nuclear medicine physician and radiologist on presence of local recurrent or metastatic lesions

SECONDARY OUTCOMES:
Differences in detection rates between 68Ga- and 18F-PSMA tracers | baseline
  Comparison of detection rates between the two radioisotopes based on consensus scoring
Differences in detection rates after radical treatment between whole-body PET/CT with and without PET/MR | baseline
  Comparison of number of present local recurrent or metastatic lesions
Number of equivocal findings with and without addition of PET/MR to the whole-body PET/CT | baseline
  Comparison of the number of local recurrent and metastatic lesions scored as equivocal
Detection rates of the combined PET/MR and PET/CT protocol compared with MRI-only. | baseline
  Comparison of detection rates using MRI only compared to the detection rates based on consensus decision using the combined PET/MR and PET/CT protocol
Detection rate dependency on prostate specific antigen (PSA) level and kinetics at time of imaging in addition to Gleason score and stage of primary cancer | baseline
  Detection rates stratified according to PSA levels, kinetics and Gleason score
Inter-reader variability for interpretation of the PSMA PET/CT and PET/MR | baseline
  Retrospective re-evaluation of images at minimum three sites
Detection of differences in image quality between participating centra | baseline
  Image quality will be scored on a 5-point Likert Scale by a nuclear medicine physician and radiologist and compared between the centra
Sensitivity and specificity of the standardized whole-body PET/CT and targeted PET/MR protocol for detection of recurrence based on long-term clinical follow-up | baseline images and long term follow-up
  A reference standard based on evidence from histopathology, clinical follow-up and follow-up imaging will be established using criteria defining presence and absence of local recurrent and metastatic disease
Head to head comparison of uptake patterns of 68Ga- and 18F-PSMA | baseline
  A selected subset of patients will be invited for a second imaging session.
Evaluation of locoregional PET-uptake according to primary radical treatment | baseline
  Comparison of locoregional PET-uptake in patients treated with primary radiotherapy versus primary prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, phd, Study Director — NTNU, Fac of Med and Health Sci, Dept of Circulation and Medical Imaging; Edmund Søvik, md phd, Study Director — St Olavs Hospital, Dept of Radiology and Nuclear Medicine
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
We will consider to openly share a completely anonymized dataset of the cohort at the end of the project